CLINICAL TRIAL: NCT00001107
Title: Invasive Fungal Infection in Liver Transplant Recipients: A Randomized Double-Blind Trial Comparing AmBisome and Fluconazole in the High Risk Group and an Observational Cohort Study in the Low Risk
Brief Title: Comparison of Two Treatments to Prevent Invasive Fungal Infections in Patients Who Have Received Liver Transplants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: DMID 98-014; MSG #44
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Candidiasis
MeSH Terms: conditions — Candidiasis | interventions — Fluconazole; liposomal amphotericin B

INTERVENTIONS:
Drug: Fluconazole
Drug: AmBisome

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of 2 treatments to prevent invasive fungal infections (IFI), which are infections caused by yeasts and molds that are common in patients with weak immune systems or transplant patients. AmBisome, a new treatment, will be compared to fluconazole, the traditional treatment for fungal infections caused by the yeast Candida. Treatment will only be given to liver transplant patients who are found to be at high risk for IFI. Liver transplant patients who are at low risk for IFI will be monitored but will receive no study medication.

IFIs are found mainly in a high risk group of liver transplant patients, and are not common in those with low risk. If IFI preventive therapy is focused on the high risk group, there may be a lesser chance of Candida becoming resistant (able to grow despite the presence of drugs used to kill it). Treating only the high risk group will also save money.

DETAILED DESCRIPTION:
If you are in the high risk group you will be assigned randomly (like tossing a coin) to receive either AmBisome or fluconazole. If you are in the low risk group, you will not receive any treatment. Both groups will be monitored for IFIs. The study will last for 100 days following your liver transplant.

ELIGIBILITY:
Inclusion Criteria:

You may be eligible for this study if you:

* Have had a liver transplant within 5 days of enrollment and agree to receive tacrolimus.

Exclusion Criteria:

You will not be eligible for this study if you:

* Are HIV-positive.
* Have a history of invasive fungal infection.
* Have received antifungal agents within 14 days prior to your liver transplant.
* Are allergic to azoles, amphotericin B, or tacrolimus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Ellen Bradley, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Hadley S, Huckabee C, Pappas PG, Daly J, Rabkin J, Kauffman CA, Merion RM, Karchmer AW. Outcomes of antifungal prophylaxis in high-risk liver transplant recipients. Transpl Infect Dis. 2009 Feb;11(1):40-8. doi: 10.1111/j.1399-3062.2008.00361.x. Epub 2008 Dec 19. PMID 19144094